CLINICAL TRIAL: NCT00711841
Title: Postpartum Dexamethasone for Women With Class I HELLP Syndrome: a Double-blind, Placebo-controled, Randomized Clinical Trial
Brief Title: Effectivity of Postpartum Dexamethasone for Women With Class I HELLP Syndrome
Acronym: COHELLP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The speed of recruitment was slower than anticipated.
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Responsible Party: Principal Investigator, Leila Katz, Obstetrical ICU obstetrical coordinator; MD , PhD, Instituto Materno Infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMIFernando Figueira
Record Dates: First submitted 2008-07-07; First posted 2008-07-09 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: HELLP Syndrome
Keywords: HELLP syndrome; dexamethasone; postpartum period; class I HELLP syndrome
MeSH Terms: conditions — HELLP Syndrome | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- saline solution (Placebo Comparator): Placebo (saline solution), 2 mL, intravenous, every 12 hours, for 48 hours
  Interventions: Drug: dexamethasone; Drug: Placebo
- Dexamethasone (Active Comparator): Dexamethasone, 10mg (2mL), intravenous, every 12 hours, for 48 hours
  Interventions: Drug: dexamethasone

INTERVENTIONS:
Drug: dexamethasone — Dexamethasone, 10mg (2mL), intravenous, every 12 hours, for 48 hours
  Arms: saline solution
Drug: Placebo — Saline solution, 2 mL, intravenous, every 12 hours, for 48 hours
  Arms: saline solution
Drug: dexamethasone — dexamethasone, 10mg, 2 mL, intravenous solution, every 12 hours , for 48 hours
  Arms: Dexamethasone

SUMMARY:
Corticotherapy accelerates maternal postpartum recovery in women with class I HELLP syndrome. The benefit of faster and better recovery would be observed in fewer complications, less utilization of blood products and shorter hospital stay.

DETAILED DESCRIPTION:
Patients with Class I HELLP Syndrome will be recruited for use os dexamethasone or placebo in the puerperium. Effects such as clinical course (blood pressure and diureses), laboratorial behaviour and complications will be compared. Duration of hospitalization will also be accessed.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women with Class I HELLP syndrome

Exclusion Criteria:

* Chronic users of corticosteroids
* Patients with chronic conditions affecting the laboratory parameters involved in the HELLP syndrome
* Women who had received antenatal corticosteroids to treat HELLP syndrome were excluded

Ages: 13 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2011-07; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
severe maternal morbidity | postpartum
  42 days after delivery

SECONDARY OUTCOMES:
hospital stay duration | postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Leila Katz, pHD, Principal Investigator — IMIP
Locations (1):
- Instituto Materno Infantil Prof. Fernando Figueira, Recife, Pernambuco, Brazil

REFERENCES:
- [Derived] Katz L, Amorim M, Souza JP, Haddad SM, Cecatti JG; COHELLP Study Group. COHELLP: collaborative randomized controlled trial on corticosteroids in HELLP syndrome. Reprod Health. 2013 May 22;10:28. doi: 10.1186/1742-4755-10-28. PMID 23697398